CLINICAL TRIAL: NCT00004356
Title: Study of Homocysteine Metabolism in Homocystinuria
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of California, San Diego (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Other Study IDs: 199/11920; UCSD-1033
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Homocystinuria
Keywords: homocystinuria; inborn errors of metabolism; rare disease
MeSH Terms: conditions — Homocystinuria; Metabolism, Inborn Errors; Rare Diseases

SUMMARY:
OBJECTIVES: I. Determine basal and postmethionine plasma homocysteine in patients with premature vascular disease, cystathionine beta-synthase (CBS) or methylenetitrahydrofolate reductase (MTHFR) deficiency, and in obligate heterozygotes for CBS or MTHFR.

II. Determine whole-body homocysteine metabolic rates with isotopically-labeled methionine.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a two-part study of homocysteine metabolism. Age-matched normal controls are entered in both parts of the study.

In first part of the study, participants are given oral methionine; baseline and postmethionine studies include amino acid quantitation, analysis of rapidly deproteinized plasma, and total plasma homocysteine.

In the second part of the study, participants (men and postmenopausal women only) undergo methionine tracer studies.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Known or suspected homocystinuria Cystathionine beta-synthase-deficient homocystinuria Obligate heterozygotes for cystathionine beta-synthase deficiency Premature vascular disease

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 1995-02; Study Completion 2000-10

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Barshop, Study Chair — University of California, San Diego

REFERENCES:
- [Background] Page T, Barshop BA, Yu A, et al.: Treatment of Lesch-Nyhan syndrome with AICAR. In: Sahota A, Tayor M, eds.: Purine and Pyrimidine Metabolism in Man VIII. Plenum Press, New York, NY: 1995, pp 353-356.